CLINICAL TRIAL: NCT05385393
Title: Functional Outcomes and the Restoration of Range of Motion After the Arthroscopic Complete Posterior Knee Capsulotomy in Patients With Extension Deficit of the Knee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Artromedical Konrad Malinowski Clinic (Other)
Responsible Party: Principal Investigator, Konrad Malinowski MD, Head of the Clinic, Artromedical Konrad Malinowski Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-pro-ar-2021
Record Dates: First submitted 2021-10-30; First posted 2022-05-23 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Knee Disease; Knee Deformity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arthroscopic posterior capsulotomy of the knee (Experimental)
  Interventions: Procedure: Arthroscopic posterior capsulotomy of the knee

INTERVENTIONS:
Procedure: Arthroscopic posterior capsulotomy of the knee — The arthroscopic posterior capsulotomy of the knee is performed according to the predefined surgical technique, which was described in detail in the following publication:
  Malinowski K, Góralczyk A, Hermanowicz K, LaPrade RF, Więcek R, Domżalski ME. Arthroscopic Complete Posterior Capsulotomy for Knee Flexion Contracture. Arthrosc Tech. 2018 Oct 15;7(11):e1135-e1139. doi: 10.1016/j.eats.2018.07.008. PMID: 30533360; PMCID: PMC6262078.

SUMMARY:
The restriction of the range of motion is one of the most frequently encountered complications after the surgical procedures of the knee. While the flexion deficit is relatively well tolerated, even the small extension deficit significantly impairs the quality of life due to the increased stress on the patellofemoral joint, functional leg length discrepancy and the subsequent mechanical overload in the hip joint, lumbar spine and contralateral knee. In the majority of cases the guided physiotherapy protocol is sufficient to restore the full range of motion. In refractory cases, the treatment consists of the thorough arthrolysis of the affected knee, aiming to excise the adhesions, osteophytes and orthopaedic implants interfering with the knee range of motion. However, as the extension deficit persists, the contracture of the knee posterior capsule may develop and the sole debridement of the knee may be insufficient. In such rare cases the treatment consists of the posterior capsulotomy of the affected joint. Traditionally, this procedure was performed through the open approach. However, with the growing indications toward the arthroscopic procedures seen in recent decades, even such salvage procedures like posterior knee capsulotomy are increasingly performed through the arthroscopic approach. The aim of this study is to assess the outcomes of the arthroscopic complete posterior capsulotomy of the knee basing on the knee range of motion and functional outcomes. The primary outcome consists of the knee extension, whereas the secondary outcomes include knee flexion, knee total range of motion, The International Knee Documentation Committee Questionnaire and the Knee injury and Osteoarthritis Outcome Score.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old,
* Symptomatic asymmetric extension deficit >3 degrees,
* Impossibility to restore the full knee extension after 6 months of guided physiotherapy.

Exclusion Criteria:

* Restoration of full knee extension after the initial knee arthrolysis,
* Active knee inflammation,
* Non-adherence of the patient to the treatment protocol.
* Contractures due to extra-articular reasons,
* Less than 6 months since the last surgical procedure affected knee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The extension of the knee | Immediately after the surgery.
  The extension of the knee will be measured with the goniometer with the patient lying supine. The hyperextension of the knee will be denoted as the negative value of knee extension.
The extension of the knee | At the 3 month of the follow-up.
  The extension of the knee will be measured with the goniometer with the patient lying supine. The hyperextension of the knee will be denoted as the negative value of knee extension.
The extension of the knee | At the 6 month of the follow-up.
  The extension of the knee will be measured with the goniometer with the patient lying supine. The hyperextension of the knee will be denoted as the negative value of knee extension.
The extension of the knee | At the 12 month of the follow-up.
  The extension of the knee will be measured with the goniometer with the patient lying supine. The hyperextension of the knee will be denoted as the negative value of knee extension.
The extension of the knee | At the 24 month of the follow-up.
  The extension of the knee will be measured with the goniometer with the patient lying supine. The hyperextension of the knee will be denoted as the negative value of knee extension.

SECONDARY OUTCOMES:
The flexion of the knee | Immediately after the surgery
  The flexion of the knee will be measured with the goniometer with the patient lying supine.
The flexion of the knee | At the 3 month of the follow-up.
  The flexion of the knee will be measured with the goniometer with the patient lying supine.
The flexion of the knee | At the 6 month of the follow-up.
  The flexion of the knee will be measured with the goniometer with the patient lying supine.
The flexion of the knee | At the 12 month of the follow-up.
  The flexion of the knee will be measured with the goniometer with the patient lying supine.
The flexion of the knee | At the 24 month of the follow-up.
  The flexion of the knee will be measured with the goniometer with the patient lying supine.
The range of motion of the knee | Immediately after the surgery
  The range of motion of the knee will be measured with the goniometer with the patient lying supine as a difference between knee flexion and knee extension.
The range of motion of the knee | At the 3 month of the follow-up.
  The range of motion of the knee will be measured with the goniometer with the patient lying supine as a difference between knee flexion and knee extension.
The range of motion of the knee | At the 6 month of the follow-up.
  The range of motion of the knee will be measured with the goniometer with the patient lying supine as a difference between knee flexion and knee extension.
The range of motion of the knee | At the 12 month of the follow-up.
  The range of motion of the knee will be measured with the goniometer with the patient lying supine as a difference between knee flexion and knee extension.
The range of motion of the knee | At the 24 month of the follow-up.
  The range of motion of the knee will be measured with the goniometer with the patient lying supine as a difference between knee flexion and knee extension.
The functional assessment with the International Knee Documentation Committee Questionnaire | Immediately after the surgery.
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the International Knee Documentation Committee Questionnaire | At the 3 month of the follow-up.
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the International Knee Documentation Committee Questionnaire | At the 6 month of the follow-up.
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the International Knee Documentation Committee Questionnaire | At the 12 month of the follow-up.
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the International Knee Documentation Committee Questionnaire | At the 24 month of the follow-up.
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score | Immediately after the surgery
  Min of 0 max of 100 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score | At the 3 month of the follow-up.
  Min of 0 max of 100 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score | At the 6 month of the follow-up.
  Min of 0 max of 100 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score | At the 12 month of the follow-up.
  Min of 0 max of 100 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score | At the 24 month of the follow-up.
  Min of 0 max of 100 points, higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Artromedical Orthopaedic Clinic, Bełchatów, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campbell TM, Trudel G. Knee Flexion Contracture Associated With a Contracture and Worse Function of the Contralateral Knee: Data From the Osteoarthritis Initiative. Arch Phys Med Rehabil. 2020 Apr;101(4):624-632. doi: 10.1016/j.apmr.2019.11.018. Epub 2020 Jan 7. PMID 31917195
- [Background] Campbell TM, Trudel G, Laneuville O. Knee flexion contractures in patients with osteoarthritis: clinical features and histologic characterization of the posterior capsule. PM R. 2015 May;7(5):466-73. doi: 10.1016/j.pmrj.2014.12.001. Epub 2014 Dec 12. PMID 25511691
- [Background] Lobenhoffer HP, Bosch U, Gerich TG. Role of posterior capsulotomy for the treatment of extension deficits of the knee. Knee Surg Sports Traumatol Arthrosc. 1996;4(4):237-41. doi: 10.1007/BF01567970. PMID 9046510
- [Background] Malinowski K, Goralczyk A, Hermanowicz K, LaPrade RF, Wiecek R, Domzalski ME. Arthroscopic Complete Posterior Capsulotomy for Knee Flexion Contracture. Arthrosc Tech. 2018 Oct 15;7(11):e1135-e1139. doi: 10.1016/j.eats.2018.07.008. eCollection 2018 Nov. PMID 30533360
- [Background] Murata Y, Takahashi K, Yamagata M, Hanaoka E, Moriya H. The knee-spine syndrome. Association between lumbar lordosis and extension of the knee. J Bone Joint Surg Br. 2003 Jan;85(1):95-9. doi: 10.1302/0301-620x.85b1.13389. PMID 12585585
- [Background] Tardy N, Thaunat M, Sonnery-Cottet B, Murphy C, Chambat P, Fayard JM. Extension deficit after ACL reconstruction: Is open posterior release a safe and efficient procedure? Knee. 2016 Jun;23(3):465-71. doi: 10.1016/j.knee.2016.01.001. Epub 2016 Feb 11. PMID 26875053
- [Derived] Malinowski K, Mostowy M, Kozlak M, Pekala PA, Kennedy NI, LaPrade RF. Complete Arthroscopic Posterior Knee Capsulotomy in Patients With Knee Extension Deficit: Preliminary Results of a Clinical Trial. Orthop J Sports Med. 2023 Dec 1;11(12):23259671231203606. doi: 10.1177/23259671231203606. eCollection 2023 Dec. PMID 38045767